CLINICAL TRIAL: NCT06391814
Title: Open-Label Individual Patient Study of Epstein-Barr Virus (EBV) Specific T-Cell Lines for the Treatment of a Lymphoproliferative Disease and Hemophagocytic Syndrome Associated With EBV
Brief Title: Donor-Derived EBV-Specific T Cells for Life Threatening EBV-lymphoma (OLIP-EBV-TCL-01-HMR01)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3579
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: EBV Associated Lymphoma
Keywords: Adoptive immunotherapy; EBV; Systemic EBV-positive T-cell lymphoma of childhood

STUDY DESIGN:
Intervention Model Description: single patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: EBV-specific T cells — Consolidative cellular immunotherapy consisting of one (or up to 4) infusion of ex vivo expanded T cells

SUMMARY:
Single-patient trial aiming to provide immunological consolidation following allogeneic stem cell transplantation to a young adult patient suffering from a systemic EBV-positive lymphoma of childhood.

DETAILED DESCRIPTION:
Following a presumed primary EBV infection, a 19 year old female patient rapidly suffered systemic inflammatory response, hemophagocytosis, multi-organ failure and evidence of EBV+ T-cell lymphoma.

The patient was aggressively treated and responded to SMILE-based chemotherapy. Once complete response was ascertained by PET imaging, the patient underwent myeloablative HLA-matched unrelated allogeneic stem cell transplantation (cyclophosphamide 60mg/Kg, total body irradiation - 12Gy with anti-thymocyte globulin). The stem cell donor had a positive serology for EBV (IgG).

The patient's EBV titer was weakly positive at the time of transplantation. A decision was made to offer consolidative treatment consisting of donor-derived ex vivo expanded EBV-reactive T cells following transplantation.

A EBV-specific T-cell line was manufactured from a portion of the cryopreserved G-CSF mobilized peripheral graft after appropriate authorizations were obtained.

The patient suffered a severe episode of intestinal graft-versus-host disease early following transplantation but received a first dose of EBV-reactive T cells (20x10e6 T cells/meter square of body surface area 5 months post-transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to provide informed consent
2. Age ≥ 18
3. Negative serum pregnancy test and use of effective contraception method.

Exclusion Criteria:

1. Administration within less than 28 days of T-cell depleting antibodies (ATG, OKT3, Campath)
2. Pregnancy
3. Any abnormal condition or laboratory result that is considered by the Principal Investigator capable of altering patient or study outcome.
4. Active uncontrolled GVHD (acute GVHD grade II-IV or progressive extensive chronic GVHD) at time of enrolment or infusion.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-04-05 (Estimated); Study Completion 2025-04-05 (Estimated)

PRIMARY OUTCOMES:
Safety of a donor-derived EBV-specific T-cell line as assessed clinically by the lack of graft-versus-host host (GVHD). | 1 year
  Evaluate the safety in terms of occurrence of graft-versus-host disease of a donor-derived allogeneic EBV-specific T-cell line generation and infusion in a patient suffering from a life-threatening EBV-related disease who received an allogeneic stem cell transplantation. Acute GVHD symptoms will be scored using MAGIC criteria using scores from 0 to IV, IV being the most severe involvement) on skin, liver and gastro-intestinal tract. Chronic GVHD symptoms will be score using the NIH consensus scale (0 to 3, 3 being the most severe) on the following organs skin, mouth, eyes, GI tract, liver, lungs, joints and fascia, and genital tract.

SECONDARY OUTCOMES:
Clinical response | 1 year
  Disease recurrence as assessed by imaging (PET scanning)
Immune reconstitution to EBV | 1 year
  Measurement of viral titers (nucleic acid testing) and peripheral blood ELISpot measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Ciusss-Emtl, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No